CLINICAL TRIAL: NCT02674269
Title: A Randomized Double-Blind, Placebo Controlled Study Evaluating the Safety and Efficacy of Intravesical Instillations of BotuGelTM, Slow Release RTGel Based Botulinum Toxin (Botox®) Formulations, in Idiopathic OAB Patients With Urinary Incontinence ("INTIMO2")
Brief Title: Safety and Efficacy Study of Intravesical Instillations of BotuGelTM, Slow Release RTGel Based Botox® Formulations, in Idiopathic OAB Patients With Urinary Incontinence ("INTIMO2")
Acronym: INTIMO2
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: UroGen's RTGelTM delivery system technology for use with neurotoxins licensed to Allergan plc before the activation of this trial.
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-OAB-03-P
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Botox; TC-3 Gel; Intravesical; UroGen Pharma; Botulinum Toxin; Urgency; OAB; Incontinence; I-QOL; KHQ; TBS; RTG
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 300 IU of BotuGelTM (60ml) (Experimental): One intravesical instillation of 300 IU of botox in 60 ml of TC-3 gel
  Interventions: Drug: 300 IU of BotuGelTM (60ml)
- 400 IU of BotuGelTM (60ml) (Experimental): One intravesical instillation of 400 IU of botox in 60 ml of TC-3 gel
  Interventions: Drug: 400 IU of BotuGelTM (60ml)
- TC-3 Gel (Placebo Comparator): One intravesical instillation of 60 ml TC-3 gel
  Interventions: Device: TC-3 Gel

INTERVENTIONS:
Drug: 300 IU of BotuGelTM (60ml) — One intravesical instillation of 300 IU of botox in 60 ml of TC-3 gel
  Other Names: BotuGelTM 300
  Arms: 300 IU of BotuGelTM (60ml)
Drug: 400 IU of BotuGelTM (60ml) — One intravesical instillation of 400 IU of botox in 60 ml of TC-3 gel
  Other Names: BotuGelTM 400
  Arms: 400 IU of BotuGelTM (60ml)
Device: TC-3 Gel — Intravesical instillation of 60 ml TC-3 gel
  Arms: TC-3 Gel

SUMMARY:
The study will investigate the safety and efficacy of UroGen's TC-3 Gel for sustained release of Botulinum Toxin A (BTX) in urinary bladder in patients with idiopathic overactive bladder.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a syndrome, defined by the International Continence Society (ICS), as the presence of "urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of a urinary tract infection (UTI) or other obvious pathology." This study will evaluate a new of mode of treatment, with intravesical bladder instillation with Botox® mixed with TC-3 that may bypass the drawbacks of the current bladder injection treatment mode in OAB patients. Additionally it will provide preliminary safety and efficacy data that may serve as a basis for a larger study exploring safety and efficacy aspects of this new mode of treatment.

50 patients will be randomized in a horse race fashion in a ~2:2:1 ratio. The patients will be screened for up to 3 weeks prior to treatment.

The patients will be requested to stop their OAB medications 7 days prior to treatment visit. 20 patients will receive one instillation of 300U of BotuGel (60ml), 20 patients will receive one instillation of 400U of BotuGel (60ml) and 10 patients will receive one instillation of 60 ml RTGel-TC-3 Gel (Placebo), all patients will be followed up for safety and efficacy endpoints until 6 weeks post instillation.

ELIGIBILITY:
Main Inclusion Criteria:

* Female patient 18 to 75 years old diagnosed with idiopathic OAB.
* Patient has symptoms of OAB for ≥ 3 months prior to screening.
* Patient is a non-responder to pharmacologic therapy or has intolerable side effects or is not compliant to the treatment.
* On screening three-day voiding diary- Patient has a frequency of at least 8 micturitions per 24 hours & Total of ≥3 urgency urinary incontinence (UUI) episodes.
* Patient is willing and able to initiate self catheterization post-treatment, if required.
* Patients has PVR ≤100 ml. Patient with a single PVR of >100 ml and followed by two consecutive PVR measurements of <100 ml may be included in the study).

Main Exclusion Criteria:

* Patient currently uses CIC or indwelling catheter to manage their urinary incontinence
* Patient who has clinically significant Bladder Outlet Obstruction (BOO).
* Patient with active urinary tract infection.
* OAB due to any known neurological reason.
* Patient with 24-hour total urine volume voided greater than 3,000 ml as measured at screening visit.
* Predominance of stress incontinence in the opinion of the investigator, determined by patient history.
* Use of anticholinergics or other medications or therapies to treat symptoms of OAB within 7 days of screening.
* Patient with prior botulinum toxin therapy of any serotype within 12 weeks for any indication.
* Patient with prior use of Botulinum toxin therapy of any serotype for any urological condition.
* Patient with previous pelvic radiation therapy.
* Patient had been treated for two or more UTIs within last 6 months or use of prophylactic antibiotics to prevent chronic UTIs.
* ANY condition identified which may cause overactive bladder symptoms

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Estimated); Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Urinary retention | 6 weeks
  Urinary retention events defined as a PVR >200 and <350 ml with patient reported symptoms that in the investigator's opinion require initiation of CIC, or PVR≥350 regardless of symptoms.
Urinary tract infection (UTI) events | 6 weeks
  Urinary tract infection (UTI) events*
  *Asymptomatic bacteruria will not be considered UTI and will be reported as separate AEs.
Post-void residual (PVR) | 6 weeks
  PVR-Change from baseline in PVR as measured by bladder ultrasonography at week 4 post instillation
Adverse events | 6 weeks
  Adverse events during and post instillation procedure.

SECONDARY OUTCOMES:
3-day voiding Diary | Week 4 and 6 post-instillation
  3-day voiding Diary
  * Change from baseline in number of Urgency episodes and Urinary Incontinence episodes/24h
  * Change from baseline in number of voids/24h
  * Change from baseline in number of nocturnal voids per night (Based on individual patient's night and day hours)
  * Change from baseline in Mean volume voided per micturition/24h
Kings Health Questionnaire (KHQ score) comparing to baseline | Week 4 and 6 post-instillation
  KHQ score comparing to baseline
Incontinence Quality of Life Questionnaire (I-QOL) | Week 4 and 6 post-instillation
  I-QOL score comparing to baseline
Treatment Benefit Scale (TBS) | Week 4 and 6 post-instillation
  Proportion of patients who had positive treatment response per Treatment Benefit Scale (TBS)
Comparison of resulted delta scores between the treatment arms and Placebo | Week 4 and 6 post-instillation

CONTACTS AND LOCATIONS:
Overall Officials: Ifat Klein, PhD, Study Director — iklein@urogen.com
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba